CLINICAL TRIAL: NCT03144856
Title: Phase II Study of Apatinib as Second Line Therapy in Patients With Advanced Refractory Biliary Tract Cancer
Brief Title: Apatinib as Second Line Therapy in Patients With Advanced Refractory Biliary Tract Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Fenghua Wang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Apatinib_BTC
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Biliary Tract Cancer
Keywords: Biliary Tract Cancer; Second line thrapy; Apatinib
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: Apatinib single agent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib group (Experimental): Apatinib 500mg, po, QD, every 4 weeks.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib 500mg, po, qd, every 4 weeks.

SUMMARY:
This study is designed to see whether Apatinib is effective in treating patients with advanced refractory biliary tract cancers.

DETAILED DESCRIPTION:
Biliary tract cancers (BTC) includes cholangiocarcinoma and gallbladder carcinoma (GBC). The systematic treatment based on gemcitabine plus cisplatin is recommended as the current standard chemotherapy for unresectable or metastatic BTC. There is no standard recommendation for second line therapy.

Apatinib is a tyrosine kinase inhibitor targeting vascular endothelial growth factor receptor 2(VEGFR-2).

This study was conducted to assess the efficacy and safety of Apatinib in patients with advanced refractory BTC who had received first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Must have histologically or cytologically documented carcinoma primary to the intra- or extra-hepatic biliary system or gall bladder with clinical and/or radiologic evidence of unresectable, locally advanced or metastatic disease.
2. Patients with ampullary carcinoma are not eligible.
3. Must have failed or are intolerant to one line of systemic treatment but no more than 2 prior lines of systemic chemotherapy for advanced BTC. Patients who received adjuvant chemotherapy and had evidence of disease recurrence within 6 months of completion of the adjuvant treatment are also eligible. If the patient received adjuvant treatment and had disease recurrence after 6 months, patients will only be eligible after failing or having intolerance to one line of systemic chemotherapy used to treat the disease recurrence.
4. Age between 18 and 75 years old
5. Eastern Cooperative Oncology Group (ECOG) Performance Status Assessment of 0 or 1.
6. Must have radiographic measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
7. Life expectancy of at least 12 weeks (3 months).
8. For patients who have received prior radiation, cryotherapy, radiofrequency ablation, therasphere, ethanol injection, transarterial chemoembolization (TACE) or photodynamic therapy, the following criteria must be met: 28 days have elapsed since that therapy; Lesions that have not been treated with local therapy must be present and measureable.
9. Must be able to understand and be willing to sign the written informed consent form. Must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other study requirements.
10. All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v4.0 Grade 1 or less at the time of signing the Informed Consent Form (ICF) except for alopecia.
11. Adequate bone marrow, liver and liver function.
12. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug.
13. Men and women of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 3 months after the last dose of study drug.

Exclusion Criteria:

1. Pregnant or lactating women;
2. History of other malignancies except cured basal cell carcinoma of skin and carcinoma insitu of uterine cervix;
3. Uncontrolled hypertension;
4. Intercurrence with one of the following: coronary artery disease, arrhythmia and heart failure;
5. Urine protein>grade 1;
6. Any factors that influence the usage of oral administration;
7. Patients with a clear tendency of gastrointestinal bleeding;
8. Abnormal coagulation function(INR≥1.5, APTT≥1.5 ULN);
9. Abuse of alcohol or drugs;
10. Less than 4 weeks from the last clinical trial;
11. Prior treatment with antivascular endothelial growth factor or the other anti angiogenesis therapy;
12. Active central nervous system (CNS). If CNS metastases are treated and potential participants are at neurologic baseline for at least 2 weeks prior to enrollment, they will be eligible but will need a Brain MRI prior to enrollment. 13. Disability of serious uncontrolled intercurrence infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 1 year
  the time from randomize to progression or death; RECIST guidelines were used to define all responses after patients had received every 4 weeks of therapy

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 2 years
  Defined as the time from randomize to death
Disease control rate(DCR) | Approximately 1 year
  Defined as the rate of complete response , partial response and stable disease according to RECIST guidelines
Quality of life(QoL) | Approximately 1 year
  As measured by the European Organization for Research and Treatment of Cancer questionnaire (EORTC QLQ C30)
Safety (incidence of adverse events) | Approximately 1 year
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Rui-Hua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Foshan people's Hospital, Foshan, Guangdong
  - Cancer center of Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No